CLINICAL TRIAL: NCT00851214
Title: Assessments of Early Hemodynamics in Emergency Department Patients and Evaluation of Trends and Variability in Prediction of Life-saving Interventions
Brief Title: Use of Non Invasive Hemodynamic Cardiovascular Monitoring to Evaluate Emergency Department Patients
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: BMEYE, Amsterdam The Netherlands (Unknown)
Responsible Party: Richard M. Nowak MD, Henry Ford Hospital
Other Study IDs: HFH DEM 001
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2009-03

CONDITIONS: COPD; Congestive Heart Failure; Trauma; Sepsis; Stroke
Keywords: Non-invasive hemodynamic monitoring; Emergency Department patients; trauma with an ISS>15; Non-invasive continuous hemodynamic monitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Wounds and Injuries; Sepsis; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Acute CHF/COPD: Patients presenting with shortness of breath secondary to acute exacerbation of CHF/COPD
  Interventions: Device: NexfinHD Monitor
- Acute Trauma: Acute trauma patients with a trauma ISS>15
  Interventions: Device: NexfinHD Monitor
- Sepsis: Patients presenting with a suspicion of acute sepsis (fever, tachycardia, tachypnea)
  Interventions: Device: NexfinHD Monitor
- Stroke: Patients presenting with symptoms and signs of acute stroke (thrombotic or hemorrhagic)
  Interventions: Device: NexfinHD Monitor

INTERVENTIONS:
Device: NexfinHD Monitor — Finger cuff device (NexfinHD Monitor, BMEYE, Amsterdam) that can measure hemodynamics on a beat to beat basis and that can be easily applied to acutely ill individuals.
  Other Names: Transcient Ischemic Attack

SUMMARY:
This study is an observational prospective pilot trial that utilizes finger cuff non invasive hemodynamic monitoring (NexfinHD Monitor) to assess 4 different groups (CHF/COPD, Trauma, Sepsis, Stroke) of patients on arrival to the Emergency Department and to document the changes seen in these hemodynamics with acute therapies.

DETAILED DESCRIPTION:
There has been little very early (after Emergency Department presentation) hemodynamic monitoring of acutely ill or injured patients secondary to the lack of non invasive technologies that could be reliably applied to this patient population.Thus all assessments of hemodynamics have been made by physicians on clinical information including intermittent pulse and blood pressure measurements. It is not known what the underlying continuous cardiac output, systemic vascular resistance, etc are in these patients and how these change with current Emergency Medicine therapeutic interventions. Currently there is available a finger cuff devise (NexfinHD Monitor, BMEYE, Amsterdam) that can measure these hemodynamics on a beat to beat basis and that can be easily applied to acutely ill individuals. This prospective pilot study of 48 patients (4 groups of 12 each) will document the hemodynamics of patients on arrival and continuously for 2 hours, blinded to the treating physician. Treating physicians will be asked to estimate these hemodynamic parameters at various time points. The study will characterize the hemodynamics of patients, compare them to the estimates of treating physicians and determine whether they predict the need for life saving interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute CHF/COPD (n=12)
* Patients with acute trauma and a trauma ISS>15 (n=12)
* Patients with acute sepsis (n=12)
* Patients with acute stroke (n=12)

Exclusion Criteria:

* Patients in cardiopulmonary arrest
* patients with STEMI
* Patients with known peripheral vascular disease
* Pregnant patients
* Age<18
* Excessively agitated patients
* Interference with current standard of acre

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely ill or injured Emergency Department patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To elucidate the hemodynamics of the cohort of four different groups of patients in the early hours of their presentation | Emergency Department (ED) arrival to 2 hours

SECONDARY OUTCOMES:
Comparison of clinical estimation of hemodynamics and values estimated by the NexfinHD on arrival and for up to 6 hours | ED arrival to 6 hours
To compare if abnormal hemodynamics as measured by the NexfinHD and clinical assessment after arrival to the ED in the 4 groups predicts life saving interventions within 2 hours | ED arrival to 2 hours
To calculate short term hemodynamic variability parameters and their prediction of life saving interventions within 2 hours and subjective/objective estimation of clinical improvement | ED arrival to 2 hours
Estimation of bias and precision of the non invasive hemodynamic trends in unselected patient group by assessing the validity of measurements with invasive measurements if used | ED arrival to 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Nowak, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital Emergency Department, Detroit, Michigan, United States

REFERENCES:
- [Derived] Nowak RM, Sen A, Garcia AJ, Wilkie H, Yang JJ, Nowak MR, Moyer ML. Noninvasive continuous or intermittent blood pressure and heart rate patient monitoring in the ED. Am J Emerg Med. 2011 Sep;29(7):782-9. doi: 10.1016/j.ajem.2011.05.014. Epub 2011 Jul 29. PMID 21802881